CLINICAL TRIAL: NCT04606056
Title: A Single Center Observational Study- Incidence and Risk Factors of Acute Kidney Injury After Intravenous Contrast Enhanced Computed Tomography Scans
Brief Title: Risk of Acute Kidney Injury After Intravenous Contrast Computed Tomography Scans
Status: Active, not recruiting | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005-00046
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury; Contrast-induced Nephropathy
Keywords: Intravenous; contrast; acute kidney injury; computer tomography
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent contrast enhanced CT scans

SUMMARY:
Intravenous iodinated contrast media is commonly used to enhance diagnostic yield of computer tomography (CT) scans in clinical medicine. However, the perceived risk of contrast-induced nephropathy (CIN) frequently limits its use. While CIN is often self-limiting, it can cause significant morbidity by prolonging admissions and rendering an at-risk individual dialysis dependent. CIN has long been observed and described in clinical studies. There is ample data on CIN after administration of intraarterial contrast, but evidence is less compelling when it comes to intravenous contrast. Increasing studies have called into question the actual risk of intravenous contrast media. Expert panels are suggesting that the risk could have been overstated, leading to contrast being withheld when indicated. There is paucity of local data on this particular issue. More real world data on the actual incidence and risk factors of AKI will be helpful to clinicians.

The investigators plan to conduct a single center, retrospective study, to determine the incidence and risk factors of post contrast AKI in contrast enhanced CT scans.

DETAILED DESCRIPTION:
A single center, retrospective study will be conducted, looking into all patients who had contrast-enhanced CT scans done in a specified time period. Serum creatinine at baseline and at 48-72 hours post-contrast of the participants will be compared to determine presence of post contrast AKI (PC-AKI). Data on the participants' demographics, comorbidities, laboratory results and use of nephrotoxins will also be captured and analysed.

The primary objective of this study is to determine the incidence of AKI after intravenous contrast administration for contrast enhanced CT scans (CECT). The secondary objective is to identify risk factors of PC-AKI and possibly come up with a risk stratification system that can be utilized in clinical practice. The investigators hypothesize that there is significant risk of acute kidney injury after intravenous contrast media administration, but it lower than that in the setting of intraarterial contrast; and that risk factors of AKI may include: pre existing chronic kidney disease, diabetes, hypertension, proteinuria, use of nephrotoxins, age, increased dose of contrast.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent one or more CT scan in CGH in the stipulated study period
2. CT scan done as an inpatient or outpatient of CGH
3. Serum creatinine available less than 6 months before scan
4. Serum creatinine available within 1 week after scan

Exclusion Criteria:

1. Age 12 or below
2. Dialysis dependent before scan (dialysis related charge code applied 24 months before scan)
3. Baseline serum creatinine not available
4. Post scan serum creatinine not available

Ages: 13 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient of an acute care hospital with clinical indications for contrast enchanced CT scans, meeting inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | 31 May 2020 to 30 June 2020
  within 1 week after contrast exposure

CONTACTS AND LOCATIONS:
Overall Officials: Chang Yin Chionh, FASN, Study Chair — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davenport MS, Khalatbari S, Dillman JR, Cohan RH, Caoili EM, Ellis JH. Contrast material-induced nephrotoxicity and intravenous low-osmolality iodinated contrast material. Radiology. 2013 Apr;267(1):94-105. doi: 10.1148/radiol.12121394. Epub 2013 Jan 29. PMID 23360737
- [Background] McDonald JS, McDonald RJ, Carter RE, Katzberg RW, Kallmes DF, Williamson EE. Risk of intravenous contrast material-mediated acute kidney injury: a propensity score-matched study stratified by baseline-estimated glomerular filtration rate. Radiology. 2014 Apr;271(1):65-73. doi: 10.1148/radiol.13130775. Epub 2014 Jan 16. PMID 24475854
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Leow KS, Wu YW, Tan CH. Renal-related adverse effects of intravenous contrast media in computed tomography. Singapore Med J. 2015 Apr;56(4):186-93. doi: 10.11622/smedj.2015057. PMID 25917468
- [Background] Davenport MS, Khalatbari S, Cohan RH, Dillman JR, Myles JD, Ellis JH. Contrast material-induced nephrotoxicity and intravenous low-osmolality iodinated contrast material: risk stratification by using estimated glomerular filtration rate. Radiology. 2013 Sep;268(3):719-28. doi: 10.1148/radiol.13122276. Epub 2013 Apr 11. PMID 23579046
- [Background] Davenport MS, Perazella MA, Yee J, Dillman JR, Fine D, McDonald RJ, Rodby RA, Wang CL, Weinreb JC. Use of Intravenous Iodinated Contrast Media in Patients With Kidney Disease: Consensus Statements from the American College of Radiology and the National Kidney Foundation. Kidney Med. 2020 Jan 22;2(1):85-93. doi: 10.1016/j.xkme.2020.01.001. eCollection 2020 Jan-Feb. PMID 33015613
- [Background] Rudnick MR, Leonberg-Yoo AK, Litt HI, Cohen RM, Hilton S, Reese PP. The Controversy of Contrast-Induced Nephropathy With Intravenous Contrast: What Is the Risk? Am J Kidney Dis. 2020 Jan;75(1):105-113. doi: 10.1053/j.ajkd.2019.05.022. Epub 2019 Aug 28. PMID 31473019